CLINICAL TRIAL: NCT06788314
Title: A Single Center, Single Arm, Phase 2, Pilot Study to Investigate the Efficacy of the ACE Inhibitor Enalapril in Participants Aged 18-70 Years of Age With Painful Venous Malformations.
Brief Title: A Study of Enalapril in Treatment of Venous Malformations
Acronym: EVA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Christina Elisabeth Bjerring Opheim, Medical doctor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-510076-31-00
Record Dates: First submitted 2025-01-10; First posted 2025-01-23 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Venous Malformation; Pain; Quality of Life; Vascular Malformation
MeSH Terms: conditions — Pain; Vascular Malformations | interventions — Enalapril

STUDY DESIGN:
Intervention Model Description: Prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enalapril (Experimental)
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — Each participant will receive a dose of enalapril 5 mg once daily. If the participant doesn't have effect of the intervention after 3 months, the dose of enalapril will be increased to 10 mg daily, if the tolerance of enalapril is good. Lack of effect will be defined as unchanged or increased NRS score.
  Treatment duration will be 12 months.

SUMMARY:
The goal of this clinical trial is to explore if enalapril can be used to treat painful venous malformations. The main question it aims to answer are:

- Can enalapril reduce pain and volume of the malformation and increase quality of life in patients with painful venous malformations?

Participants will:

Receive a dose of enalapril 5 mg once daily. If it doesn't have effect the dose of enalapril will be increased to 10 mg daily after 3 months.

The treatment duration will be 12 months, with an additional follow-up of 12 months.

The visit frequency will be after 1, 3, 6,9 and 12 months and then a follow up visit at 18 and 24 months.

Approximately 15 participants will be screened to achieve minimum 10 enrolled participants.

DETAILED DESCRIPTION:
Venous malformations are congenital defects of vasculature and may be disabling for patients throughout life, mostly because of disfigurement and pain. The patients remain challenging to treat as standard of care like sclerotherapy and compression garment is often inadequate in relieving the symptoms.

A chance observation has given reason to believe that enalapril may have the potential to reduce pain and volume in venous malformations. A young man with a symptomatic intramuscular venous malformation of the upper limp, and hypertension was treated with an angiotensin-converting enzyme (ACE) inhibitor (enalapril). After 8 months of treatment, it was registered a considerable volume reduction of the malformation and a reduction in pain.

Studies have reported that embryonic stem cell-like subpopulations in venous malformations express components of the renin-anigotensin system (RAS).

It has been hypothesized that such primitive cells could be a novel therapeutic target by manipulation of the RAS using ACE-inhibitors.

The aim of the study is to explore if the chance observation of reduced pain and volume of a venous malformation after enalapril treatment is a coincidence, or if enalapril may play a future role in the treatment of venous malformations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with venous malformations verified by clinical examination, ultrasound and anatomic MRI with contrast. The venous malformation should have well defined borders and the volume should be measurable on MRI. Diagnosis of venous malformation shall be object for consensus in a multidisciplinary team meeting.
2. Patients must experience pain from the malformation. Pain is defined as local pain in the malformation, and the participant must have pain that according to the patient inhibits daily activity or pain during nighttime that interferes with sleep. The symptoms has to reduces quality of life. NRS inclusion criteria is greater or equal to 4.
3. Participant must be 18 to 70 years of age inclusive, at the time of signing the informed consent.
4. Negative urine pregnancy test in females with childbearing potential. A woman is considered of childbearing potential i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.
5. Woman of childbearing potential (WOCBP) must use highly effective contraception measures while on study medicine and for up to 2 weeks past treatment:

   * Combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation.
   * Progestogen-only hormonal contraception associated with inhibition of ovulation Intrauterine device (IUS) Intrauterine hormone-releasing system (IUS) Bilateral tubal occlusion Vasectomized partner Sexual abstinence (controlled with regular questioning by PI)
6. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF). They must also be capable of answer adequately questionnaires regarding quality of life. Since the questionnaire are validated in Norwegian and English they also should control one of this language.

Exclusion Criteria:

1. Diffuse VM with no defined borders.
2. Known diabetes because of the risk of hypoglycemia.
3. Impaired liver function (INR > 1,5 or aminotransferases > 3 times upper limit of normal
4. Use of mTOR-inhibitor, racekadotril, sacubitril/valsartan, ramipril or vildagliptin is contraindicated because of an elevated risk of angioedema
5. Use of angiotensin-II receptor antagonist or alsikiren (direct renin inhibitor) is contraindicated because of increased risk of hypotension, hyperkalemia, and impaired renal function.
6. Impaired cardiac function and clinically significant cardiac disease including aorta- and mitral valve stenosis and hypertrophic cardiomyopathy.
7. Lactose intolerance, total lactase deficiency or glucose-galactose malabsorption because Enalapril contains lactose.
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the ACE-inhibitor (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea > grade 2, malabsorption syndrome, or small bowel resection.)
9. Hypersensitivity to the active substance or any of the excipients listed in section 6.1 of the SmPC of enalpril or to other ACE-inhibitors.
10. Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicated participation in the clinical study.
11. Known renal artery stenosis.
12. Patients with a history of angioneurotic edema related to previous treatment with ACE-inhibitors and patients with Hereditary or ideopatic anigioneurotic edema.
13. Contraindications for MRI (cardiac pacemaker or defibrillator, intracranial clips, cochlear implants or other metallic foreign bodies, claustrophobia.
14. BMI> 30
15. Impaired kidney function (eGFR< 50)
16. Pregnant or lactating woman
17. Any condition that in the view of the investigator would suggest that the patient is unable to compley with the study protocol and procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
To explore the change of venous malformation related pain | From baseline and to the end of treatment at 12 months.
  Changes in NRS (Numeric rating scale). NRS is an analogue scale with numbers from 0-10, where 0 represents no pain and 10 represents the worst imaginable pain.

SECONDARY OUTCOMES:
To explore volume change of the venous malformation | From baseline to the end of treatment at 12 months.
  Volume will be assessed by MRI. To estimate the volume of the venous malformation the area of the malformation on multiple adjacent MRI slices will be added and multiplied by the slice thickness. The volume change at follow-up imaging is calculated according to this formula: (Volume at baseline - volume at follow up)/ (volume at baseline) x 100 = percentage volume change.
To explore change in quality of life in patients with venous malformations | From baseline to the end of treatment at 12 months.
  Quality of life, will be assessed by the SF-36 (Short Form) questionnaire. The SF-36 consists of 36 questions measuring quality of life in 4 mental domains and 4 physical domains, supplying general information about life quality. The score of the SF-36 ranging from 0-100. Higher score ranging better health status.
To explore change in quality of life in patients with venous malformations | From baseline to the end of treatment at 12 months.
  Quality of life, will be assessed by the OVAMA score (Outcome measures for vascular malformations).
  The OVAMA score is a disease specific patient-reported-outcome-measures consisting of 23 questions measuring quality of live with a general symptom scale with 6 items, a head and neck symptom scale with 8 items, and an appearance scale with 9 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway, Norway

IPD SHARING:
Plan to Share IPD: No
The data protection officer in Norway does not allow it.

REFERENCES:
- [Background] Siljee S, Keane E, Marsh R, Brasch HD, Tan ST, Itinteang T. Expression of the Components of the Renin-Angiotensin System in Venous Malformation. Front Surg. 2016 May 3;3:24. doi: 10.3389/fsurg.2016.00024. eCollection 2016. PMID 27200356
- [Background] Tan EMS, Siljee SD, Brasch HD, Enriquez S, Tan ST, Itinteang T. Embryonic Stem Cell-Like Subpopulations in Venous Malformation. Front Med (Lausanne). 2017 Oct 4;4:162. doi: 10.3389/fmed.2017.00162. eCollection 2017. PMID 29046873
- [Background] Tan EMS, Brasch HD, Davis PF, Itinteang T, Tan ST. Embryonic Stem Cell-like Population within Venous Malformation Expresses the Renin-Angiotensin System. Plast Reconstr Surg Glob Open. 2019 Apr 2;7(4):e2170. doi: 10.1097/GOX.0000000000002170. eCollection 2019 Apr. PMID 31321175
- [Background] Berger S, Bjark TH, Midtvedt K, Andersen R. Regression of a venous malformation during angiotensin-converting enzyme inhibitor treatment for hypertension. J Vasc Surg Cases Innov Tech. 2022 Sep 17;8(4):657-659. doi: 10.1016/j.jvscit.2022.09.004. eCollection 2022 Dec. PMID 36262918